CLINICAL TRIAL: NCT02605668
Title: Providing Tools for Effective Care and Treatment of Anxiety Disorders (AD): Outcomes, Mediators and Moderators of Enhanced Extinction
Brief Title: Providing Tools for Effective Care and Treatment of Anxiety Disorders
Acronym: PROTECT-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Ruhr University of Bochum (Other); University Medicine Greifswald (Other); Charite University, Berlin, Germany (Other); University of Wuerzburg (Other); Philipps University Marburg (Other); Wuerzburg University Hospital (Other); Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01EE1402A; DRKS00008743 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2015-08-24; First posted 2015-11-16 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Panic Disorder; Agoraphobia; Specific Phobias; Social Anxiety Disorder
Keywords: Anxiety Disorders; Extinction Learning; Optimized Extinction; Behavioral Therapy; Massed Confrontation; Social Anxiety Disorder; Specific Phobia; Panic Disorder; Agoraphobia
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Phobia, Specific; Phobia, Social; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensified Psychological Intervention (Experimental): Intensified psychological intervention (Cognitive Behavioral Therapy), based on optimized extinction learning
  Interventions: Behavioral: Intensified psychological intervention
- Treatment As Usual (Active Comparator): Standard intervention (Cognitive Behavioral Therapy) without optimized extinction learning
  Interventions: Behavioral: Standard intervention

INTERVENTIONS:
Behavioral: Intensified psychological intervention — 12 sessions of Cognitive Behavioral Therapy a 100 minutes, over the course of 6 weeks (2 sessions per week/week 1 and 2, 3 sessions per week/week 3 und 4, 1 session per week/week 5 and 6)
  Arms: Intensified Psychological Intervention
Behavioral: Standard intervention — 12 sessions of Cognitive Behavioral Therapy a 100 minutes, over the course of 10 weeks (2 sessions per week/week 1 and 2, 1 session per week/week 3 to 10)
  Arms: Treatment As Usual

SUMMARY:
PROTECT-AD is a cognitive behavioral treatment study involving highly qualified psychotherapeutic centers at seven German universities.

It is our goal to further investigate and optimize existing effective treatments of anxiety disorders. In order to achieve this, the investigators want to investigate the effect of extinction learning in an "intensified" psychological intervention on treatment outcome in adults and children with anxiety disorders.

The intensified psychological intervention is characterized by a higher number of exposure trials over a short time period. In the control condition the exposure trials take place in a weekly interval, analog to standard care.

DETAILED DESCRIPTION:
Novel preclinical research evidence suggests extinction learning as the core mechanism of action of exposure-based therapies and provides according strategies to improve the effectiveness of treatment by optimized extinction. A translational research agenda is suggested to examine whether enhanced extinction learning components derived from preclinical research, applied within an "intensified" exposure-based treatment, improves outcomes. In a multicenter randomized clinical trial, linked to mechanistic subprojects, the investigators test in n=620 patients with primary AD allowing for comorbidity whether intensified psychological interventions based on augmented extinction learning (IPI) result in faster, stronger and more persistent outcomes on subjective, clinical, behavioral, physiological and neural indices as compared to an, otherwise identical, standard research treatment without explicit enhanced extinction (TAU). The investigators hypothesize that (a) enhanced extinction elements (IPI) will result in higher effect sizes, faster recovery, (b) more pronounced changes in an array of systems, including elements of extinction learning and in objective behavioral measures assessed in intersession exposure trials. The investigators also examine moderators of outcome (i.e. type of diagnosis, comorbidity) and explore whether IPI is associated with lower health care costs.

ELIGIBILITY:
Inclusion Criteria:

* age 15 - 70 years
* one or more of the following DSM-IV/5 anxiety disorders: Panic Disorder, Agoraphobia, Social Anxiety Disorder, Specific Phobia
* HAMA - Score > 18
* CGI - Score > 3
* Can attend therapy regularly (with or without support)
* Informed Consent

Exclusion Criteria:

* Every reason the protocol may not be upheld (e.g. planned hospitalization within study time frame, planning to move away, etc.)
* Current suicidal tendency
* DSM-5 Bipolar Disorder
* DSM-5 Psychotic Disorder
* DSM-5 Borderline Personality Disorder
* Current treatment of other mental disorder (drugs, psychotherapy)
* Current Alcohol, Benzodiazepine or other Substance Use Disorders
* Severe medical illness/condition (every serious physical illness, including cardiovascular, kidney, endocrinological and neurological conditions, Hepatitis or other clinical findings that suggest a severe illness and may affect participation in the study)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
change in somatic and psychic anxiety symptoms | assessed three times: Baseline, Post (1 week after end of therapy) and Follow up (6 months after end of therapy)
  Anxiety symptoms are assessed using the clinician-rated Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A for the HAMA). Stronger, faster and more persistent reduction of anxiety symptoms in the IPI group than in the TAU group is expected.

SECONDARY OUTCOMES:
change in severity of the anxiety disorder | assessed five times: Baseline, therapy session 4 (week 2 of therapy), therapy session 11 (week 5 to week 9 of therapy), Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  Severity of the anxiety disorder is assessed by the clinician-rated Clinical Global Impression Scale (CGI). It is anchored for anxiety disorders.
change in categorial diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV/5) | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  categorical diagnoses are assessed using a German version of the Composite International Diagnostic Interview (CIDI).
change in screened anxiety symptoms | assessed fivetimes: Baseline, therapy session 4 (week 2 of therapy), therapy session 11 (week 5 to week 9 of therapy), Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  The DSM-5 cross-cutting symptom measure for anxiety disorders ("Cross-D") is used as a brief screener for anxiety symptoms.
change in depressive symptoms | assessed fivetimes: Baseline, therapy session 4 (week 2 of therapy), therapy session 11 (week 5 to week 9 of therapy), Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  depressive symptoms are assessed using the Beck Depression Inventory (BDI-II)
change in anxiety sensitivity | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  anxiety sensitivity is assessed using the Anxiety sensitivity inventory (ASI)
change in panic and agoraphobic symptoms | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  panic and agoraphobic symptoms are assessed using the Panic and agoraphobia scale (PAS)
change in agoraphobic avoidance | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  agoraphobic avoidance is assessed using the Mobility Inventory (MI)
change in symptoms of Generalized Anxiety Disorder | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  symptoms of generalized anxiety disorder (GAD)are assessed using the GAD-7
change in social anxiety | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  social anxiety is assessed using the Liebowitz Social Anxiety Scale (LSAS)
change in Specific Phobia symptoms | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  symptoms of specific phobia are assessed using an adapted version of the DSM-5 dimensional scale for specific phobias
change in disability | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  Disability is assessed using the 12-item version of the World Health Organization Disability Schedule (WHODAS 2.0)
change in quality of life | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  Quality of life is assessed using the EuroQol five-dimensional measure for quality of life (EQ5D)
change in psychopathological symptoms | assessed seven times: Baseline, therapy sessions 2 (week 1 of therapy), 4 (week 2), 7 (week 3 to 5), 10 (week 4 to 8), 11 (week 5 to 9), 12 (week 6 to 10) Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  psychopathological symptoms are assessed using the Brief Symptom Inventory (BSI), a short form of the Symptom Checklist 90 (SCL-90). At Baseline, Post and Follow Up, the 53 item Version is used, during therapy the 18 item version is used
change in agoraphobic cognitions | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  agoraphobic cognitions are assessed using the Agoraphobic Cognitions Questionnaire (ACQ)
fear of body sensations | assessed three times: Baseline, Post (1 week after end of therapy) and Follow Up (6 months after end of therapy)
  fear of body sensations is assessed using the Body Sensations Questionnaire (BSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Ulrich Wittchen, Ph.D., Principal Investigator — Technische Universität Dresden
Locations (1):
- Technische Universität Dresden, Institute of Clinical Psychology and Psychotherapy, Dresden, Saxony, Germany

REFERENCES:
- [Background] Heinig I, Pittig A, Richter J, Hummel K, Alt I, Dickhover K, Gamer J, Hollandt M, Koelkebeck K, Maenz A, Tennie S, Totzeck C, Yang Y, Arolt V, Deckert J, Domschke K, Fydrich T, Hamm A, Hoyer J, Kircher T, Lueken U, Margraf J, Neudeck P, Pauli P, Rief W, Schneider S, Straube B, Strohle A, Wittchen HU. Optimizing exposure-based CBT for anxiety disorders via enhanced extinction: Design and methods of a multicentre randomized clinical trial. Int J Methods Psychiatr Res. 2017 Jun;26(2):e1560. doi: 10.1002/mpr.1560. Epub 2017 Mar 21. PMID 28322476

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02605668/Prot_SAP_000.pdf